CLINICAL TRIAL: NCT02059707
Title: LARIAT RS: An Observational Study of the Performance and Safety of the LARIAT RS Suture Delivery Device
Brief Title: LARIAT RS: An Observational Study of the Performance and Safety of the LARIAT RS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AtriCure, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: RS-003 V1.0_30Oct2012
Record Dates: First submitted 2014-02-06; First posted 2014-02-11 (Estimated); Last update posted 2020-01-09 (Actual); Status verified 2017-03

CONDITIONS: Atrial Appendage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LAA exclusion procedure (Experimental): LAA exclusion with the LARIAT RS Suture Delivery Device
  Interventions: Device: LARIAT RS Suture Delivery Device

INTERVENTIONS:
Device: LARIAT RS Suture Delivery Device — LARIAT RS Suture Delivery Device

SUMMARY:
The objective is to assess the effectiveness of permanent exclusion of the LAA with the LARIAT RS Suture Delivery Device and accessories in AF patients.

DETAILED DESCRIPTION:
Prospective, observational, single-center, non-randomized study of a stand-alone procedure for the exclusion of the LAA with the LARIAT RS in patients with atrial fibrillation. Completed LAA exclusion will be assessed by TEE.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 21 years
2. Diagnosed non-valvular atrial fibrillation
3. Current CHADS2 score ≥ 2
4. Poor candidate (e.g., contraindicated, labile INR, non-compliant, etc.) for anticoagulation (e.g., warfarin, dabigatran, apixaban, and rivaroxaban)
5. Life expectancy of ≥ 1 year
6. Willing and able to provide written informed consent
7. Willing and able to come to and comply with scheduled follow-up visits

Exclusion Criteria:

1. Previous cardiac surgery involving opening of pericardium (e.g., CABG, heart transplantation, valve surgery)
2. Prosthetic heart valve or ring in any position
3. Current NYHA Class IV heart failure symptoms
4. Current right heart failure
5. Myocardial infarction or unstable angina within last 3 months
6. Current cardiogenic shock or hemodynamic instability
7. Current symptomatic carotid disease
8. Need for an intra-aortic balloon pump or intravenous inotropes
9. Embolic stroke or transient ischemic attack (TIA) within the last 30 days.
10. Current diagnosis of active systemic infection
11. Need for emergent cardiac surgery (e.g., cardiogenic shock)
12. Current renal failure requiring dialysis
13. Current clinical evidence of cirrhosis
14. Any history of thoracic radiation
15. Current use of long term treatment with steroids, not including intermittent use of inhaled steroids for respiratory diseases
16. Diagnosed autoimmune disease known to be associated with pericarditis (i.e., specific connective tissue disorders)
17. Any history of pericarditis
18. Pectus excavatum (clinically defined by treating physician)
19. Severe scoliosis
20. Pregnancy or desire to get pregnant within the next 12 months.
21. LVEF < 30%
22. Current participation in a clinical investigation that involves an active treatment arm.
23. Mental impairment or other conditions, which may not allow patient to understand the nature, significance and scope of the study
24. Any other criteria, which would make the patient unsuitable to participate in this study as determined by clinical site Principal Investigator (e.g., an uncontrolled drug and/or alcohol addiction)

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2014-01; Primary Completion 2014-12 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Percent of subjects with complete exclusion | 90 days
  To assess the rate of complete exclusion of the LAA measured by color duplex TEE at 4 time points: Acute (i.e., immediately after LAA exclusion procedure), 1 day, 1 month, and 3 month.

SECONDARY OUTCOMES:
Secondary Exploratory objectives of procedural success and device-related complication rates | 3 month
  * The rate of procedural success
  * The rate of complications related to the use of the LARIAT RS and accessories

CONTACTS AND LOCATIONS:
Locations (1):
- Jagiellonian University (John Paul II) Hospilal, Krakow, Poland